CLINICAL TRIAL: NCT06432257
Title: The Effect of the Application of Head Mounted Magnifying Glasses on Postoperative PTH Changes in Thyroid Surgery
Status: Completed | Type: Observational
Sponsor: Shandong Provincial Hospital (Other Government)
Collaborators: Shandong University (Other)
Responsible Party: Principal Investigator, Guojun Wu, Principal Investigator, Shandong Provincial Hospital
Other Study IDs: NO.SWYX2024-280
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer; PTH; Head mounted magnifying glass
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Using the head mounted magnifying glass: This study was divided into an experimental group and a control group based on whether a head mounted magnifying glass was used, with the main calculation indicator being changes in PTH levels before and after surgery.
  Interventions: Device: head mounted magnifying glass assistance

INTERVENTIONS:
Device: head mounted magnifying glass assistance — When performing thyroid surgery for patients in the experimental group, the surgeon uses a head mounted magnifying glass for assistance

SUMMARY:
This study collected data on open thyroidectomy patients admitted to the Breast and Thyroid Surgery Department of Shandong Provincial Hospital from January 2020 to December 2023 by reviewing medical records. This study was divided into an experimental group and a control group based on whether a head mounted magnifying glass was used, with the main calculation indicator being changes in PTH levels before and after surgery. This study investigated whether the application of head mounted magnifying glasses had an impact on preoperative and postoperative changes in PTH levels through inter group and self pre - and post control, in order to verify the practical effectiveness of head mounted magnifying glasses in thyroid surgery and provide reasonable suggestions for the selection of subsequent surgical treatment methods.

DETAILED DESCRIPTION:
In thyroid surgery, changes in postoperative parathyroid hormone (PTH) levels have a significant impact on the patient's recovery and long-term health status. Parathyroid hormone is responsible for regulating blood calcium levels, and its dysfunction can cause serious electrolyte imbalance and metabolic problems. In the process of thyroid surgery, especially in total thyroidectomy, protecting the function of the parathyroid gland is an important operation. The diameter of the parathyroid gland is small and similar to the morphology of lymph nodes, making it susceptible to damage during surgery. Although traditional magnification tools such as surgical microscopes have certain effects, their operation is complex and their adaptability to surgical scenes is limited.

In recent years, as an emerging magnifying tool, head mounted magnifying glasses have been increasingly used in thyroid surgery due to their portability, ease of operation, and providing a larger field of view. Wearing a head mounted magnifying glass can not only improve the clarity of vision during surgery, increase the recognition rate of parathyroid glands and nerves, but also reduce the risk of parathyroid injury by improving surgical accuracy, thereby more effectively maintaining the stability of postoperative PTH levels. In addition, the use of head mounted magnifying glasses can reduce surgical time, intraoperative uncertainty, and the risk of postoperative complications.

This study systematically evaluates the changes in PTH levels before and after surgery to verify the practical effectiveness of head mounted magnifying glasses in thyroid surgery, and further explores the effectiveness of parathyroid gland protection strategies, optimizing surgical techniques, and improving patient surgical safety and postoperative quality of life. In addition, the results of this study also have guiding significance for the innovation and improvement of surgical instruments, which may promote the development of related technologies and equipment, and thus promote their application in a wider range of surgical fields.

ELIGIBILITY:
Inclusion Criteria:

* All cases were the first to undergo open thyroidectomy surgery.
* All clinical data and research materials of the cases are complete.
* All cases underwent thyroid function examination before and after surgery.
* All cases in the experimental group were treated with a head mounted magnifying glass during surgery.

Exclusion Criteria:

* Except for cases of recurrence.
* Cases with incomplete clinical data and research materials are excluded.
* Cases that have not undergone thyroid function tests before and after surgery are excluded.
* Excluding cases of secondary surgery.
* Excluding cases in the experimental group who did not use a head mounted magnifying glass during surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study collected patients who underwent open thyroidectomy surgery at the Breast and Thyroid Surgery Department of Shandong Provincial Hospital from January 2020 to December 2023. All patients included in the study had complete clinical and research data, with approximately 2000 participants.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
PTH level | 4 weeks
  To verify the practical effectiveness of wearing a magnifying glass in thyroid surgery by examining changes in PTH levels before and after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong provincial hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
The data are not publicly available due to privacy and ethical restrictions.